CLINICAL TRIAL: NCT03621228
Title: A Pilot Study of an Interactive Digital Technology (MindfulGarden) in Treatment of Hyperactive Delirium in a Hospital Setting
Brief Title: MindfulGarden in Treatment of Hyperactive Delirium in a Hospital Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Gloria Gutman, Professor Emerita, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MindfulGarden-H-Pilot
Record Dates: First submitted 2018-07-27; First posted 2018-08-08 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Hyperactive Delirium
Keywords: Delirium; Hyperactive; Aggression; Anxiety; Digital therapy
MeSH Terms: conditions — Delirium; Spasm; Aggression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MindfulGarden (Experimental): Standard care + exposure to an interactive digital device
  Interventions: Device: MindfulGarden
- Control (No Intervention): Standard care only

INTERVENTIONS:
Device: MindfulGarden — MindfulGarden (MG) is an interactive digital technology that combines use of a smart television with sensors to intelligently generate content based on patient voice and gesture input, triggering a multi-layered visual 'garden' on-screen to arrest and de-escalate anxiety and aggression in treatment of hospitalized elderly diagnosed with hyperactive delirium.
  Arms: MindfulGarden

SUMMARY:
This pilot study is designed to address feasibility for a larger randomized control clinical study that will determine the efficacy of exposure to the MindfulGarden - an interactive digital technology - in reducing hyperactive delirium in hospitalized older adults.

DETAILED DESCRIPTION:
The primary objective of the study is to establish whether the key components necessary for conducting a full randomized control study in the future, such as recruitment, consent, randomization, and treatment processes are working well and all function together. As a secondary objective, the investigators will determine trends in patients exposed to MindfulGarden (MG), for example:

1. At the first and second administration of the Confusion Assessment Method - short form (CAM) after admission to a medical ward are there more, the same or fewer patients in the intervention group than in the control group whose CAM scores change from positive to negative?
2. During the first 24 hours after admission to a medical ward, did fewer, the same, or a greater number of patients in the intervention than in the control group experience significant events/alerts (e.g. aggressive/violent behaviours, falls, code white)?
3. During the first 24 hours after admission to a medical ward, were fewer, the same, or a greater number of patients in the intervention than in the control group administered psychotropic drugs (e.g. haloperidol, risperidone, quetiapine, lorazepam)? were more, the same, or fewer administered sleeping aids (e.g. trazodone, melatonin)?
4. During the first 24 hours after admission to a medical ward, were fewer, the same, or a greater number of patients in the intervention than in the control group physically restrained?
5. Was mean length of stay from time of admission to a medical ward until discharge due to death, return to place of residence before admission or to a different place of residence longer, the same or shorter in the intervention than in the control group?
6. Were there more, the same or fewer deaths or discharges to a higher level of care (e.g. to assisted living, to a complex care facility in patients who previously lived at home) in the intervention than the control group?

Additionally, to the extent that movement and vocalization are reflective of anxiety, agitation and/or aggression (i.e. responsive behaviours) the investigators also want to determine whether there is a correlation between changes in these as recorded by the MG and any of the indicators listed in 1-6 above.

ELIGIBILITY:
Inclusion Criteria:

- All patients aged 65 years or older admitted to the Emergency Department who have a diagnosis of hyperactive delirium as defined by the short CAM

Exclusion Criteria:

* Patients with severe vision impairment or who are legally blind
* Patients for whom a bed in a medical ward was not available within 12 hours of a diagnosis of hyperactive delirium (i.e. who remained in the Emergency Department more than 12 hours)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | Number enrolled within 12 hours of admission to Emergency Department
  Number of participants approached and their rate of consent

SECONDARY OUTCOMES:
Estimate the potential effect size | 24-hour period following transfer from Emergency Department
  MG association with reducing delirium duration as measured CAM - short
Adverse Outcomes (number of patients with aggressive/violent behaviours, falls, code white) | 24-hour period following transfer from Emergency Department
  Assess from patients medical chart
Psychotropic Drug Consumption | 24-hour period following transfer from Emergency Department
  Assess from patient's medical chart
Application of Physical Restraints | 24-hour period following transfer from Emergency Department
  Assess from patient's medical chart
Length of Stay | Date of study enrolment through to discharge from hospital, or date of study enrolment up to 30 days
  Assess from patient's medical chart

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Gutman, Principal Investigator — Simon Fraser University

IPD SHARING:
Plan to Share IPD: No